CLINICAL TRIAL: NCT06592638
Title: A Phase 1 Dose Escalation Study of the Tolerability, Safety, Efficacy and Pharmacokinetics of ZG006 in Patients With Small Cell Lung Cancer
Brief Title: A Phase 1 Dose Escalation Study of ZG006 in Patients With Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZG006US001
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-04

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental)
  Interventions: Drug: ZG006

INTERVENTIONS:
Drug: ZG006 — ZG006 will be administered as an intravenous (IV) infusion.

SUMMARY:
This is a multi-center, open-label, Phase 1 clinical study of ZG006 in the US for the treatment of subjects with small cell lung cancer who have failed or are intolerant to available standard treatment. During the dose escalation stage, a standard "3+3" design will be used to assess the MTD/ recommended dose for the subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* Small cell lung cancer (SCLC), who failed or intolerant to available standard treatments;
* Tissue sample positive for DLL3 expression;
* Life expectancy ≥ 3 months;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
* Female and Male patients must agree to use a reliable form of contraception during the study treatment period and for at least 6 months after the last dose of the study drug.

Exclusion Criteria:

* Patients having received any of the following treatments:

  * Chemotherapy, biotherapy, endocrine therapy (except for hormone replacement), and biological targeted medicines ≤ 4 weeks before the study entry. Local palliative radiotherapy and a small molecule targeted therapy ≤ 2 weeks (or 5 half-lives, whichever is longer) before the study entry;
  * Systemic immunosuppressive medications, such as corticosteroid (doses > 10 mg/day prednisone or equivalent dose) within 14 days prior to the study entry;
  * Use of any vaccines against viral infections (COVID-19, influenza, varicella, etc.) within 4 weeks of study entry;
* Patients received any blood transfusion, EPO, G-CSF, albumin infusion and renal replacement therapy within 14 days prior to study entry;
* A history of severe, life-threatening immune-mediated adverse events or infusion-related reactions during previous anti-tumor immunotherapy, including events that led to permanent discontinuation of treatment;
* Active infection (such as acute bacterial infection, tuberculosis, active hepatitis B/C, active syphilis, or active human immunodeficiency virus infection);
* Known allergy to other mAbs or any antibody excipients; the history of a severe allergic reaction, anaphylactoid or other hypersensitivity reactions to humanized antibodies or fusion proteins;
* A female who is pregnant or nursing;
* Patients were deemed unsuitable for participating in the study by the investigator for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicity (DLT) | Up to 28 days
  An event is considered to be a DLT if the event occurs within the first 28 days of treatment and meets the dose-limiting toxicity criteria
Maximum Tolerated Dose (MTD) of ZG006 | Approximately 2 years
Determine the Recommended Phase 2 Dose (RP2D) | Approximately 2 years
Number of participants with adverse events (AEs) | Approximately 2 years
  The types and frequencies of adverse events (AEs) evaluated according to the National Cancer Institute Common Terminology Criteria for adverse events (NCI-CTCAE) version 5.0
Number of participants with serious adverse events (SAEs) | Approximately 2 years
Incidence of abnormal laboratory results | Approximately 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | Approximately 2 years
  ORR is defined as the percentage of participants achieving a confirmed complete response (CR) or partial response (PR) based on RECIST 1.1 criteria.
Duration of response (DOR) | Approximately 2 years
  DOR is defined as the time from first evidence of response (CR or PR per RECIST 1.1) to earlier date of disease progression or death due to any cause
Disease control rate (DCR) | Approximately 2 years
Maximum plasma concentration (Cmax) of ZG006 | Approximately 2 years
Time to peak concentration (Tmax) | Approximately 2 years
AUC from time zero to the last quantifiable concentration after dosing (AUC[0-t]) of ZG006 | Approximately 2 years
Terminal phase half-life (t1/2) of ZG006 | Approximately 2 years
Detection of anti-drug antibodies (ADA) | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Zelgen Site 105, Orange, California
  - Zelgen Site 102, Plantation, Florida
  - Zelgen Site 103, Lexington, Kentucky
  - Zelgen Site 101, Canton, Ohio
  - Zelgen Site 104, Cleveland, Ohio
  - Zelgen Site 106, Houston, Texas